CLINICAL TRIAL: NCT00268775
Title: Implementation Strategies Aimed at a Simple Patient-directed Intervention to Reduce Long-term Use of Benzodiazepines in Dutch Community Pharmacies
Brief Title: Implementation Strategies for a Simple Intervention to Reduce Longterm Benzodiazepine Use in Dutch Community Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Zorgverzekeraar CZ (Other); Scientific Institute for Dutch Pharmacists, The Netherlands (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: WOK/WINAp/CZ-01
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Benzodiazepines Therapeutic Use
Keywords: community pharmacy services; patient care; outcome assessment; benzodiazepines therapeutic use

INTERVENTIONS:
Behavioral: training and follow-up of pharmacists
Behavioral: patient-directed discontinuation letter

SUMMARY:
The purpose of this study is to compare the effect of two implementation strategies for a simple patient-directed intervention to reduce long-term benzodiazepine use in Dutch community pharmacies.

DETAILED DESCRIPTION:
In Dutch community pharmacies many projects have been undertaken in the field of pharmaceutical care, with mixed results. It is not yet clear which elements exactly contribute to the success of these projects and to implementation of pharmaceutical care.

One of the subjects to which attention is paid in community pharmacies, is the undesirable long-term use of benzodiazepines. Treatment methods for discontinuation of long-term benzodiazepine use have been studied rather extensively. A simple patient-directed discontinuation letter proved to be effective in several studies.

Comparison: a minimal intervention group (pharmacists carrying out the intervention guided by a manual only) compared to a maximal intervention group (pharmacists receiving a manual, a training aimed at better cooperation and communication with family practitioners and some support in the management of the project).

ELIGIBILITY:
Inclusion Criteria:

* benzodiazepine use for more than 3 months in the last 12 months AND for more than 60 days in the last 2 months

Exclusion Criteria:

* treatment by psychiatrist, treatment of alcohol- or drug misuse, psychotic episodes in history, epilepsy, terminal disease, not mastering the Dutch language, individual criteria used by the family practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
percentage of general practitioners that reviewed and returned the list of longterm users.
percentage of letters sent by the pharmacists in the four months after receiving the manual.
percentage of long-term benzodiazepine users that managed to quit or significantly reduce their use in months 0-3, 4-6 and 10-12 after receiving the letter.

SECONDARY OUTCOMES:
evaluation of the implementation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Peter G de Smet, PhD, Principal Investigator — Scientific Institute for Dutch Pharmacists, The Netherlands; Michel Wensing, PhD, Study Director — Centre for Quality of Care Research Nijmegen
Locations (90):
- Netherlands (90):
  - Apotheek Schellekens, 's-Hertogenbosch
  - Apotheek Cleij, 's-Hertogenbosch
  - Apotheek Empel, 's-Hertogenbosch
  - Apotheek Asten, Asten
  - Apotheek Bakel-Milheeze, Bakel
  - Kring-apotheek Bergeyk, Bergeijk
  - Apotheek Berlicum, Berlicum
  - Lloyds Apotheek van Kollenburg, Best
  - Apotheek de Schakel, Best
  - Apotheek Heivelden, Best
  - Apotheek Blanckenburgh, Beuningen
  - Apotheek Bladel, Bladel
  - Apotheek Bocholtz, Bocholtz
  - Apotheek van de Wouw, Brunssum
  - Apotheek Budel, Budel
  - Apotheek in 't Groen, Deurne
  - Apotheek Koolen-Motké, Deurne
  - Apotheek de Schelde, Deurne
  - Apotheek Druten, Druten
  - Apotheek de Kempen, Eersel
  - Apotheek Elsloo, Elsloo
  - Apotheek Ewijk, Ewijk
  - Apotheek Eygelshoven, Eygelshoven
  - Lloyds Apotheek Geldrop, Geldrop
  - Apotheek het Frans Brugske, Gemert
  - Apotheek Lindner, Gemert
  - Apotheek de Duivenakker, Gennep
  - Apotheek Gennep, Gennep
  - Apotheek de Pijlers, Goes
  - Zeeuwse Apotheek, Goes
  - Apotheek de Goese Polder, Goes
  - Apotheek Groesbeek, Groesbeek
  - Linde apotheek, Hapert
  - Apotheek Heeswijk-Dinther, Heeswijk-Dinther
  - Apotheek Tendijck, Helmond
  - Service Apotheek de Bus, Helmond
  - Service apotheek Vondellaan, Helmond
  - Apotheek de Luifel, Helmond
  - Apotheek Brouwhuis, Helmond
  - Kring-apotheek de Rijpel, Helmond
  - Lloyds Apotheek Herkenbosch, Herkenbosch
  - Apotheek Hegtermans, Herten
  - Apotheek Herten-Merum, Herten
  - apotheek Kerkrade-centrum, Kerkrade
  - Apotheek Schonefeld, Kerkrade
  - Apotheek Bleijerheide, Kerkrade
  - Apotheek Medische Centrum West Kerkrade, Kerkrade
  - Apotheek Terwinselen, Kerkrade
  - Apotheek Waubach, Landgraaf
  - Apotheek Landgraaf, Landgraaf
  - Apotheek MC Putstraat, Landgraaf
  - Apotheek Schaesberg, Landgraaf
  - Apotheek Nieuwenhagen, Landgraaf
  - Apotheek Maarheeze, Maarheeze
  - Apotheek Craveld, Maasbracht
  - Apotheek Maasbracht, Maasbracht
  - Service apotheek Malden, Malden
  - Apotheek Maasdorpen, Meerlo
  - Lloyds Apotheek de Roerstreek, Melick
  - Apotheek Ringeling, Middelburg
  - Apotheek Hummelen, Middelburg
  - Apotheek Stromenwijk 't Zand, Middelburg
  - Apotheek Welsinge, Middelburg
  - Apotheek Dauwendaele, Middelburg
  - Apotheek van der Ploeg, Nijmegen
  - Kring-apotheek Beckers, Nijmegen
  - Apotheek Souburg, Oost-Souburg
  - Lloyds Apotheek Postert, Posterholt
  - Apotheek Reusel, Reusel
  - Lloyds Apotheek Clemens-Haan, Roermond
  - Reinald apotheek, Roermond
  - Apotheek Hendrickx-Maasniel, Roermond
  - Lloyds Apotheek Donderberg, Roermond
  - Apotheek Roermond Zuid, Roermond
  - Apotheek Rosmalen-Walschot, Rosmalen
  - Apotheek Rosmalen, Rosmalen
  - apotheek Simpelveld-Bocholtz, Simpelveld
  - Apotheek Hopveld, Sint-Michielsgestel
  - Apotheek de Baandert, Sittard
  - Wandelbos Apotheek, Tilburg
  - Apotheek de Belleman, Valkenswaard
  - Apotheek Valkenswaard, Valkenswaard
  - Apotheek Vlaslant, Valkenswaard
  - Apotheek Dommeldal, Valkenswaard
  - apotheek 't Zuid, Veghel
  - Veldhovense Apotheek, Veldhoven
  - Apotheek Zonderwijk, Veldhoven
  - Apotheek van Poppel, Wijchen
  - Apotheek Dr. H. Kilian, Wijchen
  - Apotheek Wijchen-Zuid, Wijchen

REFERENCES:
- [Background] Odedina FT, Hepler CD, Segal R, Miller D. The Pharmacists' Implementation of Pharmaceutical Care (PIPC) model. Pharm Res. 1997 Feb;14(2):135-44. doi: 10.1023/a:1012032223328. PMID 9090699
- [Background] Anderson GM, Lexchin J. Strategies for improving prescribing practice. CMAJ. 1996 Apr 1;154(7):1013-7. PMID 8625021
- [Background] Grimshaw JM, Shirran L, Thomas R, Mowatt G, Fraser C, Bero L, Grilli R, Harvey E, Oxman A, O'Brien MA. Changing provider behavior: an overview of systematic reviews of interventions. Med Care. 2001 Aug;39(8 Suppl 2):II2-45. PMID 11583120
- [Background] Collins TM, Mott DA, Bigelow WE, Zimmerman DR. A controlled letter intervention to change prescribing behavior: results of a dual-targeted approach. Health Serv Res. 1997 Oct;32(4):471-89. PMID 9327814
- [Background] Muijrers PE, Knottnerus JA, Sijbrandij J, Janknegt R, Grol RP. Changing relationships: attitudes and opinions of general practitioners and pharmacists regarding the role of the community pharmacist. Pharm World Sci. 2003 Oct;25(5):235-41. doi: 10.1023/a:1025872907411. PMID 14584231
- [Background] Zitman FG, Couvee JE. Chronic benzodiazepine use in general practice patients with depression: an evaluation of controlled treatment and taper-off: report on behalf of the Dutch Chronic Benzodiazepine Working Group. Br J Psychiatry. 2001 Apr;178:317-24. doi: 10.1192/bjp.178.4.317. PMID 11282810
- [Background] Vorma H, Naukkarinen H, Sarna S, Kuoppasalmi K. Long-term outcome after benzodiazepine withdrawal treatment in subjects with complicated dependence. Drug Alcohol Depend. 2003 Jun 5;70(3):309-14. doi: 10.1016/s0376-8716(03)00014-0. PMID 12757968
- [Background] Voshaar RC, Gorgels WJ, Mol AJ, van Balkom AJ, van de Lisdonk EH, Breteler MH, van den Hoogen HJ, Zitman FG. Tapering off long-term benzodiazepine use with or without group cognitive-behavioural therapy: three-condition, randomised controlled trial. Br J Psychiatry. 2003 Jun;182:498-504. doi: 10.1192/bjp.182.6.498. PMID 12777340
- [Background] Couvee JE, Timmermans MA, Zitman FG; Dutch Chronic Benzodiazepine Working Group. The long-term outcome of a benzodiazepine discontinuation programme in depressed outpatients. J Affect Disord. 2002 Jul;70(2):133-41. doi: 10.1016/s0165-0327(01)00330-5. PMID 12117625
- [Background] Mol AJ, Oude Voshaar RC, Gorgels WJ, Breteler MH, van Balkom AJ, van de Lisdonk EH, Kan CC, Mulder J, Zitman FG. The absence of benzodiazepine craving in a general practice benzodiazepine discontinuation trial. Addict Behav. 2006 Feb;31(2):211-22. doi: 10.1016/j.addbeh.2005.04.024. Epub 2005 Jun 13. PMID 15951127
- [Background] Morin CM, Bastien C, Guay B, Radouco-Thomas M, Leblanc J, Vallieres A. Randomized clinical trial of supervised tapering and cognitive behavior therapy to facilitate benzodiazepine discontinuation in older adults with chronic insomnia. Am J Psychiatry. 2004 Feb;161(2):332-42. doi: 10.1176/appi.ajp.161.2.332. PMID 14754783
- [Background] McGregor C, Machin A, White JM. In-patient benzodiazepine withdrawal: comparison of fixed and symptom-triggered taper methods. Drug Alcohol Rev. 2003 Jun;22(2):175-80. doi: 10.1080/09595230100100615. PMID 12850904
- [Background] Gorgels WJ, Oude Voshaar RC, Mol AJ, van de Lisdonk EH, van Balkom AJ, van den Hoogen HJ, Mulder J, Breteler MH, Zitman FG. Discontinuation of long-term benzodiazepine use by sending a letter to users in family practice: a prospective controlled intervention study. Drug Alcohol Depend. 2005 Apr 4;78(1):49-56. doi: 10.1016/j.drugalcdep.2004.09.001. PMID 15769557
- [Background] Oude Voshaar RC, Gorgels WJ, Mol AJ, Couvee JE, van Balkom AJ, Zitman FG. [Treatment methods for discontinuation of long-term benzodiazepine use]. Ned Tijdschr Geneeskd. 2001 Jul 14;145(28):1347-50. Dutch. PMID 11484431
- [Background] Cormack MA, Sweeney KG, Hughes-Jones H, Foot GA. Evaluation of an easy, cost-effective strategy for cutting benzodiazepine use in general practice. Br J Gen Pract. 1994 Jan;44(378):5-8. PMID 8312045
- [Derived] van de Steeg-van Gompel CH, Wensing M, De Smet PA. Implementation of a discontinuation letter to reduce long-term benzodiazepine use--a cluster randomized trial. Drug Alcohol Depend. 2009 Jan 1;99(1-3):105-14. doi: 10.1016/j.drugalcdep.2008.07.009. Epub 2008 Sep 17. PMID 18801626